CLINICAL TRIAL: NCT02635854
Title: Study of Platelet Activation in Septic Shock Patients
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/15/7738; 15 7738 02 (Other Grant/Funding Number: University Hospital Toulouse, local funding 2015)
Record Dates: First submitted 2015-12-14; First posted 2015-12-21 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2018-08

CONDITIONS: Septic Shock
Keywords: leukocyte and platelet aggregates; platelet activation
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test group (Experimental): The test group (Septic choc group) includes 15 patients suffering from septic shock in intensive care unit.
  Interventions: Other: Septic choc group
- Control group (Other): The control group (Orthopedic surgery group) includes 15 patients recruited from the orthopedic surgical anesthesia consultation programmed for a prosthetic hip or knee pose.
  Interventions: Other: Orthopedic surgery group

INTERVENTIONS:
Other: Septic choc group — Specific platelet activation markers, circulating leukocyte-platelet aggregates will be assessed in peripheral venous blood at the admission in intensive care unit and 48 hours later for leukocyte-platelet aggregates measurements.
  Arms: Test group
Other: Orthopedic surgery group — Specific platelet activation markers, circulating leukocyte-platelet aggregates will be assessed in peripheral venous blood during the orthopedic surgical anesthesia consultation.
  Arms: Control group

SUMMARY:
Some studies have shown that antiplatelets agents could reduce organ dysfunction in septic shock in mice and human models. Platelets are actors in immunity and their activation can be complicated by tissue damage with vascular occlusions which can lead to organ dysfunction. Investigators can hypothesize an increase in platelet activation and in leukocyte-platelet aggregates in septic shock.

ELIGIBILITY:
Inclusion Criteria:

EXPERIMENTAL GROUP

* Patient who possibly gave an oral agreement to inclusion and may sign a consent once out of intensive care
* Patients hospitalized in general intensive care
* Patient hospitalized for less than 72 hours
* Patient suffering from severe sepsis, whatever their origin, with hypotension (PAs <90mmHg) despite adequate fluid resuscitation and vasoactive requiring the use of amines, with hypoperfusion and / or at least one organ dysfunction ( septic shock)
* Patient with a Sequential Organ Failure Assessment (SOFA) score> 8 (or> 2 in an organ) in the first 24 hours
* Patient enjoying a social security scheme or equivalent

CONTROL GROUP

* Signed informed consent
* Patient seen anesthesia consultation for orthopedic knee prosthesis of laying or hip with a negative balance infectious
* Patient enjoying a social security scheme or equivalent

Exclusion Criteria:

EXPERIMENTAL GROUP

* Patient on safeguarding justice, guardianship
* Patient suffering from a haematological malignancy (leukemia, lymphoma ...)
* Patient suffering from thrombocytopenia or constitutional thrombopathy
* Pregnant

CONTROL GROUP

* Patient on safeguarding justice, guardianship
* Patient with infectious positive balance (dental, urinary tract) prior to surgery
* Patient suffering from a haematological malignancy (leukemia, lymphoma ...)
* Patient suffering from thrombocytopenia or constitutional thrombopathy
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Level of platelets activation markers expression (CD62-P, antibody CD63, CD42b) | T0 at the admission in intensive care unit
  Specific platelet activation markers and circulating leukocyte-platelet aggregates will be assessed in peripheral venous blood at the admission in intensive care unit for patients in test group and during the orthopedic surgical anesthesia consultation for patients in control group.
Level of platelets activation markers expression (CD62-P, CD63, CD42b) | T48 hours after admission in intensive care unit
  Specific platelet activation markers and circulating leukocyte-platelet aggregates will be assessed in peripheral venous blood 48 hours later admission in intensive care unit only for patients in test group.

SECONDARY OUTCOMES:
Rate of leukocyte-platelet aggregates | T0 at the admission in intensive care unit
Kinetics of leukocyte-platelet aggregates formation | T0 at the admission in intensive care unit
Correlation of leukocyte-platelet aggregates rate and septic shock severity. | T0 at the admission in intensive care unit
Comparison of platelet activation in subjects treated or not with antiplatelet agents. | T0 at the admission in intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Fanny BOUNES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vardon-Bounes F, Garcia C, Piton A, Series J, Gratacap MP, Poette M, Seguin T, Crognier L, Ruiz S, Silva S, Conil JM, Minville V, Payrastre B. Evolution of platelet activation parameters during septic shock in intensive care unit. Platelets. 2022 Aug 18;33(6):918-925. doi: 10.1080/09537104.2021.2007873. Epub 2021 Dec 16. PMID 34915822